CLINICAL TRIAL: NCT07297017
Title: Naples Prognostic Score for Predicting Postoperative Delirium in the Elderly Undergoing Hip Fracture Surgeries
Brief Title: Naples Prognostic Score for Predicting Postoperative Delirium
Status: Recruiting | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gaber Ahmed, lecturer in anesthesia, Intensive Care and Pain Management, South Valley University
Other Study IDs: ِAIP003-7
Record Dates: First submitted 2025-11-25; First posted 2025-12-22 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Delirium
Keywords: POD; elderly; geriatric; NPS
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hip group: patients undergoing hip surgeries will be screened for delirium in the Post-Anesthesia Care Unit (PACU) on arrival, and once daily for the first 3 postoperative days (postoperative days 1 to 3), and on postoperative days 5 and 7.

SUMMARY:
Naples Prognostic Score (NPS) originally developed to predict outcomes in inflammatory and malignant conditions; we asked if it can effectively predict postoperative delirium (POD) in elderly patients undergoing hip surgery? NPS integrate markers such as albumin, neutrophil-to-lymphocyte ratio, and lymphocyte-to-monocyte ratio-all of which have been linked to adverse postoperative outcomes including POD.

DETAILED DESCRIPTION:
Delirium is a state of acute cerebral dysfunction that manifests as fluctuations in mental status. It is a common problem among all patients admitted to the hospital and has the potential to significantly alter patients' clinical outcomes. There are many risk factors that predispose patients to delirium including age, frailty, and preexisting comorbid conditions, as well as risk factors unique to the perioperative period, such as severity of concurrent illness, type of operation, and ICU admission after surgery (3). Postoperative delirium (POD) should be of paramount importance to providers, as multiple studies in perioperative patients have found significant associations between development of delirium within the first few days of surgery and increased length of stay, higher cost of care, increased hospital readmission rates, higher likelihood of discharge to institution, prolonged cognitive impairment and dementia, and increased mortality (4) (5) . POD occurs commonly but underdiagnosed, and is associated with worse patient outcomes.

Postoperative delirium known as a common and serious complication in elderly surgical patients, particularly after orthopedic surgeries, incidences ranging typically from 5%% up to 48%, with some reports citing rates as high as 70-80% in high-risk geriatric populations (12) . Recent literature showed a strong association between levels of nutritional parameters such as serum albumin (Alb) and lipids and an increased risk of POD (7).However, it is important to note that the prognostic power of a single marker of inflammation or nutritional index might be influenced by variations in physical conditions and the surrounding environment (8). Accordingly, the concept of using a compound indicator of nutrition state and inflammation, known as NPS, presented a novel idea for predicting POD Over the last few years, the NPS was widely used to evaluate the prognosis of cancer patients. Miyamoto et al. pointed out that the NPS was a valuable predictor for postoperative harmful outcomes in patients who underwent colorectal cancer ( CRC) and gastric cancer (GC) surgeries (9).

Because NPS combine inflammatory and nutritional indices, they may provide a more robust and easily measurable means of identifying patients at risk for POD. A preoperative tool based on these scores could enable early intervention, tailored perioperative care, and improved outcomes in this vulnerable population

ELIGIBILITY:
Inclusion Criteria:

* The elderly age≥60 years
* American Society of Anesthesiologists (ASA) classification II∼IV
* Patients undergoing hip fracture surgery
* Patients who had a complete blood sample were taken preoperatively

Exclusion Criteria:

* Patient refused to participate and consent
* Patients with a history of mild cognitive impairment (MCI), dementia, and delirium
* Ptients with known preoperative infections (pulmonary infection, urinary infection, and sepsis).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elderly patients undergoing Hip fracture surgery
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of postoperative delirium | on arrival to PACU, on postoperative day 1, 2, 3, 5, 7.
  Assessment of postoperative deliurim will be done once daily by using an established screening instrument (The Confusion Assessment Method (CAM)). A positive CAM requires both (1) Acute onset & fluctuating course AND (2) Inattention, plus (3) Disorganized thinking OR (4) Altered level of consciousness.

SECONDARY OUTCOMES:
Length of hospital stay | Directly before patients' discharge from hospital
  Determine the duration of hospital stay for geriatric hip fracture patients in our hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Qena University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No